CLINICAL TRIAL: NCT04528459
Title: Computer-Assisted Surgery for Internal Fixation of Peritrochanteric Femur Fractures: A Randomized Controlled Study
Brief Title: Computer-Assisted Fixation of Trochanteric Femur Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: ADAPT platform no longer supported
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Wakenda K. Tyler, MD, MPH, Associate Professor of Orthopedic Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAS7055
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Hip Fractures
Keywords: Peritrochanteric femur fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two treatment arms: cohort 1 will consist of patients with closed peritrochanteric femur fractures who undergo open reduction internal fixation with a Stryker© Gamma™ cephalomedullary nail using traditional fluoroscopy for insertion of the lag screw. Cohort 2 will consist of patients with closed peritrochanteric femur fractures who undergo open reduction internal fixation with a Stryker© Gamma™ cephalomedullary nail using the Stryker© ADAPT™platform to assist with insertion of the lag screw.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to treatment group allocation, as will outcomes assessors. Clinicians performing the procedures will not be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Traditional fluoroscopy (Active Comparator): Cohort 1 will consist of patients with closed peritrochanteric femur fractures who undergo open reduction internal fixation with a Stryker© Gamma™ cephalomedullary nail using traditional fluoroscopy for insertion of the lag screw (current standard of care).
  Interventions: Radiation: Traditional fluoroscopy
- Stryker© ADAPT™ platform (Experimental): Cohort 2 will consist of patients with closed peritrochanteric femur fractures who undergo open reduction internal fixation with a Stryker© Gamma™ cephalomedullary nail using the Stryker© ADAPT™platform to assist with insertion of the lag screw.
  Interventions: Device: Stryker© ADAPT™ platform

INTERVENTIONS:
Device: Stryker© ADAPT™ platform — The ADAPT system is a software platform that utilizes augmented reality to assist surgeons with implant alignment, lag screw length and positioning, and distal interlocking screw placement for cephalomedullary fixation of peritrochanteric femur fractures.
  Arms: Stryker© ADAPT™ platform
Radiation: Traditional fluoroscopy — For patients in the control group, traditional fluoroscopy will be utilized for placement of the cephalomedullary nail.
  Arms: Traditional fluoroscopy

SUMMARY:
The purpose of this study is to assess whether the Stryker© ADAPT™ augmented-reality platform can assist surgeons in optimizing placement of the lag screw component of the Stryker© Gamma™ cephalomedullary nail.

DETAILED DESCRIPTION:
This will be a prospective, randomized, single-blinded, controlled trial with two treatment cohorts. Cohort 1 will consist of patients with closed peritrochanteric femur fractures who undergo open reduction internal fixation with a Stryker© Gamma™ cephalomedullary nail using traditional fluoroscopy for insertion of the lag screw. Cohort 2 will consist of patients with closed peritrochanteric femur fractures who undergo open reduction internal fixation with a Stryker© Gamma™ cephalomedullary nail using the Stryker© ADAPT™ platform to assist with insertion of the lag screw. Patients will be blinded to treatment group allocation as will clinicians/researchers during data processing and analysis.

The primary outcome will be tip-apex distance, as measured on anteroposterior and lateral hip radiographs. Secondary outcomes will be position of the lag screw as described by Cleveland et al, operative time, fluoroscopy time, and number of Kirschner wire passes prior to final placement of the lag screw. Additionally, evidence of lag screw cutout on hip radiographs, hip range of motion relative to the contralateral hip, overall mobility, social dependency, and pain level will be assessed at 3 month, 6 month, 1 year, and 2 year follow up visits.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 18 years and older with isolated closed peritrochanteric femur fractures who are candidates for surgical fixation with a cephalomedullary nail device

Exclusion criteria:

1. Patients with open peritrochanteric femur fractures or multiple injuries (i.e., polytrauma)
2. Patients with peritrochanteric femur fractures better treated with a device other than a cephalomedullary nail, as determined by the attending orthopedic surgeon
3. Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] CLEVELAND M, BOSWORTH DM, THOMPSON FR, WILSON HJ Jr, ISHIZUKA T. A ten-year analysis of intertrochanteric fractures of the femur. J Bone Joint Surg Am. 1959 Dec;41-A:1399-408. No abstract available. PMID 13849408
- [Result] Herzog J, Wendlandt R, Hillbricht S, Burgkart R, Schulz AP. Optimising the tip-apex-distance in trochanteric femoral fracture fixation using the ADAPT-navigated technique, a longitudinal matched cohort study. Injury. 2019 Mar;50(3):744-751. doi: 10.1016/j.injury.2019.02.010. Epub 2019 Feb 13. PMID 30782395

RESULTS

PARTICIPANT FLOW:
Groups:
- Stryker© ADAPT™ Platform: Cohort 2 will consist of patients with closed peritrochanteric femur fractures who undergo open reduction internal fixation with a Stryker© Gamma™ cephalomedullary nail using the Stryker© ADAPT™ platform to assist with insertion of the lag screw.
Period: Overall Study
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.7 (12.5) | 82.0 (14.6) | 82.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Tip-apex Distance (TAD)
Description: Tip-apex distance of the lag screw in the femoral head as measured on postoperative anteroposterior and lateral x-rays
Time Frame: Immediate post-operative period
Population: Data was not collected. Participants were enrolled and randomized prior to the study termination but were not administered the study intervention.
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Lag Screw Position
Description: Lag screw position in the femoral head/neck as described by Cleveland et al. (1959)
Time Frame: Immediate postoperative period
Population: as for outcome 1
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Operative Time
Description: The amount of time required to complete the surgical procedure
Time Frame: Intraoperative period
Population: as for outcome 1
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Fluoroscopy Time
Description: The amount of fluoroscopy utilized during the surgical procedure as measured in seconds
Time Frame: Intraoperative period
Population: as for outcome 1
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: K-wire Passes
Description: The total number of K-wire passes prior to final lag screw placement
Time Frame: Intraoperative period
Population: as for outcome 1
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Evidence of Lag Screw Cut-out
Description: Evidence of lag screw cut-out as seen on postoperative hip radiographs
Time Frame: 3 months, 6 months, 1 year, and 2 years after surgery
Population: as for outcome 1
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Hip Range of Motion
Description: Postoperative range of motion of the affected hip as measured on physical examination
Time Frame: 3 months, 6 months, 1 year, and 2 years after surgery
Population: as for outcome 1
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patient Mobility and Social Dependency
Description: Postoperative patient mobility and social dependency as defined by the Harris Hip Score
Time Frame: 3 months, 6 months, 1 year, and 2 years after surgery
Population: as for outcome 1
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pain Level
Description: Postoperative pain level as defined by the visual analog scale
Time Frame: 3 months, 6 months, 1 year, and 2 years after surgery
Population: as for outcome 1
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: At time of enrollment; 1 day
Arm/Group | Traditional Fluoroscopy | Stryker© ADAPT™ Platform
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT04528459/Prot_SAP_000.pdf